CLINICAL TRIAL: NCT04996823
Title: Phase 2 Study of Axitinib + Ipilimumab in Advanced Melanoma
Brief Title: Axitinib + Ipilimumab in Advanced Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21112; 63403991 (Other: Pfizer)
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: skin cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Ipilimumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ipilimumab + Axtinib (Experimental): Participants will receive treatment with ipilimumab 3 mg/kg IV q3 weeks x 4 doses and axitinib at 5 mg by mouth twice daily. Each cycle is 3 weeks/21 days
  Interventions: Drug: Ipilimumab; Drug: Axitinib

INTERVENTIONS:
Drug: Ipilimumab — Participants will receive ipilimumab 3mg/kg IV every 3 weeks for up to 4 doses.
  Other Names: Yervoy
Drug: Axitinib — Participants will take 5 mg Axitinib twice daily by mouth for up to 35 cycles (24 months)
  Other Names: Inlyta

SUMMARY:
The goal of this clinical research study is to find out if taking axitinib with ipilimumab is effective in treating advanced melanoma.

DETAILED DESCRIPTION:
The safety and tolerability of the combination of ipilimumab and axitinib will be tested in advanced melanoma patients who are intolerable/refractory to anti-PD-1/PD-L1 therapy and have not previously received treatment with ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced/unresectable melanoma - uveal melanoma is excluded
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate bone marrow, organ function and laboratory parameters as defined in protocol.
* Patients must have adequately controlled blood pressure (<150 systolic and <100 diastolic)
* At least 1 measurable lesion - per irRECIST 1.1 criteria
* Documented disease refractory or intolerant to anti-PD-1/PD-L1 inhibitor treatment: in the metastatic setting or in the adjuvant setting if relapse on or within 6 months from end of anti-PD-1 treatment
* If BRAFV600-mutant melanoma, patients may have had prior BRAF/MEK inhibitor therapy, or intolerance to these drugs
* No limit to prior lines of treatment but prior ipilimumab not permitted
* Prior treatment-related toxicity resolved to ≤ Grade 2 or baseline
* Participants with a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Prior to first dose of study treatment, patients must be at least 2 weeks from any prior major surgery.
* Able to undergo a pre-treatment and on-treatment tumor biopsy
* Female participants of childbearing potential must have a negative serum or urine β-HCG test result. Female participants of childbearing potential and male participants must agree to use methods of contraception that are highly effective. Pregnant or breast-feeding patients are not permitted to enroll.
* Patients with brain metastases are permitted assuming that the brain metastases have been adequately treated previously. Patients with uncontrolled or symptomatic brain metastases or leptomeningeal carcinomatosis that are not stable or require corticosteroids are not permitted,
* Active autoimmune disease requiring disease-modifying therapy at the time of screening is not permitted. Replacement therapy (e.g., physiologic corticosteroid therapy) is allowed
* Participants with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 90 days prior to screening. Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment must have an undetectable HCV viral load prior to study start.

Exclusion Criteria:

* In patients with known liver cirrhosis, those with severe (Child Pugh C) hepatic impairment are excluded.
* Patients with Grade ≥3 hemorrhage within 4 weeks are excluded
* Patients with severe/unstable angina or symptomatic congestive heart failure within last 6 months are excluded
* Patients with cerebrovascular accident, transient ischemic attack within last 6 months are excluded.
* Patients with current use or anticipated need for treatment with drugs or foods that are known strong CYP3A4/5 inhibitors or strong CYP3A4/5 inducers, including their administration within 10 days prior to treatment start, are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2027-03-29 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Up to 24 months
  Overall Response Rate (ORR) defined as proportion of patients to have achieved a complete or partial response per irRECIST and RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Progression Free Survival | Up to 5 years
  Progression Free Survival (PFS) is defined as the length of time from start of study treatment to the earlier of the first documentation of disease progression or death from any cause.
Overall Survival | Up to 5 years
  Overall Survival (OS) is defined as the length of time from start of treatment to date of death from any cause.
Duration of Response | Up to 5 years
  Duration of Response is defined as the interval from the first documentation of Complete Response (CR) or Partial Response (PR) to documentation of progressive disease or death from any cause.
Clinical Benefit Rate | Up to 12 months
  Clinical Benefit Rate is defined as the proportion of patients who achieve a Complete Response (CR), Partial Response (PR) or durable Stable Disease (SD) of at least 6 months from start of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Eroglu, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States